CLINICAL TRIAL: NCT06327945
Title: Transplanting Lungs From Uncontrolled Donation After Circulatory Death: An Early Phase Clinical Trial
Brief Title: Transplanting Lungs From Uncontrolled Donation After Circulatory Death
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-00009
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lung uDCD Protocol (Experimental)
  Interventions: Device: Lung uDCD Protocol

INTERVENTIONS:
Device: Lung uDCD Protocol — The intervention is initiation of PEEP and supplemental oxygen, without requiring prior permission (e.g., for cases not having first person authorization for organ donation and organ donation for research), to offer lung donation opportunities for cases which would otherwise be ineligible in the U.S.

SUMMARY:
The study team developed an uncontrolled donation after circulatory death (uDCD) protocol that preserves lungs for just over 3 hours after death using positive end expiratory pressure (PEEP) and supplemental oxygen. The study will assess lung uDCD program safety by continuous review of operations/clinical records from each case activation and transplantation. Attrition outcomes include rates of initial and continued lung preservation, donation authorization, lung recovery, passing ex-vivo lung perfusion (EVLP) performance testing, and lung transplantation. Planned viability assessments also include macroscopic determination, radiology (X-ray), and fiber optic bronchoscopy before initiating EVLP. We expect ~50% of lungs assessed with EVLP will be transplanted to meet sustainability targets. Safety outcomes include the primary outcome, primary graft dysfunction (PGD) grade III at 72 hours, and secondarily survival one year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients waiting for lung transplants
* Willing to participate in the research study

Exclusion Criteria:

* Unable to be followed for 1 year after transplantation
* Unable to provide written informed consent to participate in the research (or designate a surrogate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Primary Graft Dysfunction (PDG) Grade III | 72 Hours Post-Transplant
  PGD is measured 72 hours after transplantation and defined according to the International Society for Heart and Lung Transplantation (ISHLT) criteria: partial pressure of arterial oxygen divided by the fraction of inspired oxygen (Pa02/FI02) < 200 mm Hg.

SECONDARY OUTCOMES:
Number of Participants who Required Normothermic Extracorporeal Membrane Oxygenation (nECMO) | 72 Hours Post-Transplant
Number of Participants who Required Normothermic Extracorporeal Membrane Oxygenation (nECMO) | 1 Year Post-Transplant
Incidence of Re-Transplantation | 1 Year Post-Transplant
Overall Survival | 72 Hours Post-Transplant
  Time from transplant to death due to any cause.
Overall Survival | 1 Year Post-Transplant
  Time from transplant to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wall, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared beginning 9 months and ending 5 years following article publication. The data will be available at a third party website. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data for any purpose will be able to access the data at a third party website.